CLINICAL TRIAL: NCT05637944
Title: ThoRAciC Trauma IntubatiON Risk Score for Blunt Trauma
Acronym: TRACTIONS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); Ospedale di Circolo e Fondazione Macchi, Varese (Unknown); Trauma Center Pisa (Unknown); Ospedale Santa Maria della Scaletta di Imola (Unknown); Azienda Ospedaliera di Perugia (Other); Ospedale Policlinico San Martino (Other); Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara (Unknown); Ospedale S. Giuseppe (Empoli) (Unknown); Pronto Soccorso Ospedale Misericordia Grosseto (Unknown); Ospedale Bufalini - Cesena (Unknown); Azienda Ospedaliero-Universitaria di Padova (Unknown); ASST Papà Giovanni XXIII Bergamo (Unknown); Pronto Soccorso e Medicina d'Urgenza Latisana (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other)
Responsible Party: Sponsor
Other Study IDs: 4860 - TRACTIONS
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Trauma Chest
Keywords: trauma; chest trauma
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intubated within day 7th: patients needing oro-tracheal intubation within day 7th from admission.
  Interventions: Procedure: oro tracheal intubation
- non intubated within day 7th: patients not requiring intubation within day 7th from admission

INTERVENTIONS:
Procedure: oro tracheal intubation — chest trauma requiring oro tracheal intubation
  Groups: intubated within day 7th

SUMMARY:
The primary objective of this study is the evaluation of risk factors associated with orotracheal intubation in blunt chest trauma patients not intubated on the field and not fulfilling the criteria for intubation based on the Glasgow Coma scale score with the building of a predictive score based on those findings taking into account the clinical, laboratory and radiologic tests performed within 6 hours from hospital admission.

DETAILED DESCRIPTION:
Multicentre, prospective, observational study. All the consecutive blunt thoracic trauma patients consecutively admitted at the participating institutions' Emergency Department (ED) will be considered for enrolment. The primary outcome measure will be the need for orotracheal intubation for primary respiratory failure lasting at least 48 hours within 7 days after trauma. The secondary outcome measures related to analgesia are: the basal analgesia protocol received during the first 7 days from ED admission and the median cumulative dose of morphine-equivalents received as rescue therapy during the first 7 days after trauma. The secondary outcome measure related to the sonographic evolution of thoracic lesions is the global and regional LUS.

ELIGIBILITY:
Inclusion Criteria:

* Blunt thoracic trauma with a documentable lesion (T-AIS ≥ 2)
* Age ≥ 18 years
* GCS > 8 at ED admission
* Total body CT scan available performed within 6 hours from ED admission

Exclusion Criteria:

* - Penetrating thoracic trauma
* Age < 18 years
* GCS <= 8 at ED admission
* Patients already intubated at ED arrival
* Do not intubate order, for any reason
* Intubation for Urgent/Emergent surgery within 24 hours from hospital arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chest trauma, blunt
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
needing for oro-tracheal intubation within day 7th from admission | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Unità Sanitaria Locale, Bologna, Italy